CLINICAL TRIAL: NCT03228524
Title: Promotion of Synaptic Plasticity With D-Aspartate to Favour Recovery Form Cerebral Damage
Brief Title: D-aspartate and Therapeutic Exercise
Acronym: DAsp&TerapEx
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Mario Stampanoni Bassi, Principal Investigator, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neuromed
Record Dates: First submitted 2017-07-12; First posted 2017-07-25 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — D-Aspartic Acid; Exercise Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Recruited patients will be randomized to receive 2660 mg D-aspartate oral dosing once daily or placebo, in addition to the conventional treatment provided by the relevant staff, for a period of 6 weeks. Patients will also be undergoing a Therapeutic Exercise Program (ET). All conventional therapies taken by patients will be recorded by the operators. Patients will be divided into two D-aspartate + ET and Placebo + ET groups and will be evaluated at zero time before starting treatment (T-0W) after 6 weeks to evaluate the effects at the end of treatment (T-6W) , And at 12 weeks (T-12W) to evaluate the maintenance of long-term effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-aspartato+ET (Experimental): Patients will be administered oral D-aspartate (2660 mg once daily) for 6 weks. Moreover, patients will receive therapeutic exercise.
  Interventions: Drug: D-Aspartate; Behavioral: Therapeutic exercise
- Placebo+ET (Placebo Comparator): Patients will be administered oral placebo for 6 weks. Moreover, patients will receive therapeutic exercise.
  Interventions: Behavioral: Therapeutic exercise; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: D-Aspartate — Patients will be randomized to receive oral D-aspartatoe (2660 mg, once daily) or placebo,as an addition to conventional therapy as indicated by physicians, for a 6 weeks period.
  Other Names: DAA, D-Aspartic acid
  Arms: D-aspartato+ET
Behavioral: Therapeutic exercise — Standard physiotherapy
  Other Names: Physiotherapy
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo+ET

SUMMARY:
An important mechanism responsible for clinical recovery after neurological damage of different types is synaptic plasticity. Nervous tissue can enhance or de-energize inter-neuronal transmission at synaptic level in a lasting way. By increasing the efficiency of synaptic transmission, through long-term potentiation (LTP), it is possible to compensate for the loss of synaptic pulses on survived neurons due to brain damage and to restore their function.

At synaptic level, LTP is mainly regulated by NMDA receptors. In animal models induction of plasticity in surviving neurons through the stimulation of NMDA receptors has been shown to limit the clinical manifestations of neuronal damage. Endogenous NMDA is synthesized by methylation of D-aspartate (Asp) by D-aspartatoartate methyltransferase . Moreover, Asp acts as a neurotransmitter capable of activating the NMDA receptor, since its biosynthesis, degradation, absorption and release occurs in the pre-synaptic neuron, and its release determines a response in Post-synaptic neurons. The expression of Asp in the SNC is very abundant during the embryonic period and in early years, whereas it is significantly reduced in adulthood.

Consistent with Asp ability of activating the NMDA receptor, recent studies have shown that oral administration of Asp increases LTP induction in mice. Preliminary studies by our group also showed an increase in LTP amplitude in subjects suffering from progressive forms of Multiple Sclerosis after 2 weeks of daily per os intake of 2660mg Asp.

It is also well known that the therapeutic exercise that characterizes a rehabilitative treatment is able to induce various benefits to the physical-functional and the cognitive-emotional spheres. In this regard, it has been extensively demonstrated how repeatedly performing a motor task can increase cortical excitability through the induction of LTP mechanisms.

Hypothesis Pharmacologically promoting the induction of cortical LTP by the intake of Asp in subjects with various types of brain damage (eg Multiple Sclerosis, Parkinson's Disease, Dementia) may favor the therapeutic effects of rehabilitative treatment.

Specific Objectives Evaluate the effects of Asp in improving the outcome of rehabilitative treatment resulting from brain damage of different origin.

DETAILED DESCRIPTION:
An important mechanism responsible for clinical recovery after neurological damage of different types is synaptic plasticity. Nervous tissue can enhance or de-energize inter-neuronal transmission at synaptic level in a lasting way. By increasing the efficiency of synaptic transmission, through long-term potentiation (LTP), it is possible to compensate for the loss of synaptic pulses on survived neurons due to brain damage and to restore their function.

At synaptic level, LTP is mainly regulated by NMDA receptors. In animal models induction of plasticity in surviving neurons through the stimulation of NMDA receptors has been shown to limit the clinical manifestations of neuronal damage. Endogenous NMDA is synthesized by methylation of D-aspartate (Asp) by D-aspartatoartate methyltransferase . Moreover, Asp acts as a neurotransmitter capable of activating the NMDA receptor, since its biosynthesis, degradation, absorption and release occurs in the pre-synaptic neuron, and its release determines a response in Post-synaptic neurons. The expression of Asp in the SNC is very abundant during the embryonic period and in early years, whereas it is significantly reduced in adulthood.

Consistent with Asp ability of activating the NMDA receptor, recent studies have shown that oral administration of Asp increases LTP induction in mice. Preliminary studies by our group also showed an increase in LTP amplitude in subjects suffering from progressive forms of Multiple Sclerosis after 2 weeks of daily per os intake of 2660mg Asp.

It is also well known that the therapeutic exercise that characterizes a rehabilitative treatment is able to induce various benefits to the physical-functional and the cognitive-emotional spheres. In this regard, it has been extensively demonstrated how repeatedly performing a motor task can increase cortical excitability through the induction of LTP mechanisms.

Hypothesis Pharmacologically promoting the induction of cortical LTP by the intake of Asp in subjects with various types of brain damage (eg Multiple Sclerosis, Parkinson's Disease, Dementia) may favor the therapeutic effects of rehabilitative treatment.

Specific Objectives A double-blind study to evaluate the effects of D-aspartate in improving the outcome of rehabilitative treatment resulting from brain damage of different origin (eg Multiple Sclerosis, Parkinson's Disease, Dementia). This will be made possible thanks to the specific skills of a multidisciplinary team of neurologists and physiatrists, healthcare professionals such as physiotherapists, occupational therapists, psychologists, speech therapists and the support of a biomedical engineer. These professional figures are already available at the UCK Neurosurgery of the IRCCS Neuromed directed by the proposer and actively collaborate to optimize the therapeutic exercise of patients with neurological damage.

Population of the study This study aims to provide preliminary data on interaction between D-aspartate and therapeutic exercise in inducing LTP cortical phenomena. The sample estimate was made by analogy after a literature analysis. In view of the quite high risk of drop out, our intention is to recruit at least 100 subjects in a population of patients with cerebral injury of various origin, coming to the neurology department of IRRCS Neuromed, Pozzilli.

Inclusion and exclusion criteria are as specified below.

Study design Double-blind prospective study, between randomized, placebo-controlled parallel groups.

Recruited patients will be randomized to receive 2660 mg D-aspartate oral dosing once daily or placebo, in addition to the conventional treatment provided by the relevant staff, for a period of 6 weeks. Patients will also be undergoing a Therapeutic Exercise Program (ET). All conventional therapies taken by patients will be recorded by the operators. Patients will be evaluated at zero time before starting treatment (T-0W) after 6 weeks to evaluate the effects at the end of treatment (T-6W) , and at 12 weeks (T-12W) to evaluate the maintenance of long-term effects. Randomization will be balanced in accordance with age, sex and schooling.

The physiotherapy and/or speech therapy approach will differ among patients considering the different types of brain damage and the different levels of disability, according to the rehabilitation unit team for each case.

Expected results The present study aims to investigate whether the association between pharmacological treatment with D-aspartate and therapeutic exercise may be more effective than just therapeutic exercise in favor of synaptic plasticity and clinical recovery under it, in patients with various forms of brain damage.

The expected result based on previous studies on mice (Errico, 2008, Errico, 2011) is that D-aspartate, promoting neuronal plasticity and acting in synergy with therapeutic exercise, strengthens the recovery of deficits in patients with various types of brain damage.

ELIGIBILITY:
This study aims to provide preliminary data on interaction between D-aspartate and therapeutic exercise in inducing LTP cortical phenomena. The sample estimate was made by analogy after a literature analysis. In view of the risk of abandonment quite high, our intention is to recruit at least 100 subjects in a population of patients with cerebral injury of various origin (such as Multiple Sclerosis, Parkinson Disease, Dementia, Skull Trauma, Stroke, Epilepsy or Other Syndromes Neurological character), related to the neurology department of IRRCS Neuromed by Pozzilli.

Inclusion criteria:

* Males or females aged between 18 and 80;
* Presence of brain damage resulting from: Multiple Sclerosis, Parkinson's Disease, Dementia, Cranial Trauma, Neurosurgery, Stroke, Epilepsy, or Other Neurological Syndromes;
* Patient's ability to adhere to the rehabilitation treatment provided for his / her clinical condition by competent personnel;
* Female subjects can not be pregnant, can not breastfeed, have been born at least three months before the beginning of the study, undertake not to schedule a pregnancy for the duration of the study;
* Patients should be able to follow protocol guidelines throughout the study;
* Patients should be able to understand the aims and risks of the study;
* Signature of informed consent, approved by our Ethics Committee.

Exclusion criteria:

* Tumors or systemic infections;
* Patients with impaired hepatic function (ALT> 3 x ULN, Alcaline Phosphatase> 2 x ULN, bilirubin tot> 2 x ULN if associated with any increase in ALT or alkaline phosphatase); Severe or moderate renal failure;
* Other contraindications or hypersensitivity to D-aspartate or its excipients;
* Patients with other pathologies which, according to the scientific officer's opinion, prevent recruitment;
* Patients unable to even partially understand and want.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Barthel's Activities of Daily Living (ADL) (O'Sullivan et al 2007) | up to 3 years
  quality of life
FIM | up to 3 years
  Functional Independence Measurement (FIM) (Chumney et al., 2010)
stroke | up to 3 years
  NIH Stroke Scale / Score (NIHSS)
disability | up to 3 years
  Expanded Disability Status Scale (EDSS) (Kurtzke, 1983)
parkinson | up to 3 years
  Unified Parkinson's Disease Rating Scale (Rammer et al. )
depression | up to 3 years
  Beck Depression Inventory (BDI) (Beck, 1972)
neuronal plasticity | up to 3 years
  Transcranial Magnetic Stimulation (TMS) will be used to evaluate the change of neuronal plasticity in a subgroup of patients who will not present contraindications to the method. The TMS uses short-lived magnetic fields and high intensity applied at the scalp level to activate the neurons of a small region of the cerebral cortex through an electromagnetic induction. When these impulses are applied repeatedly, it is possible to induce plastic modification of cortical excitability. If these changes are induced at the level of the motor cortex, they can be measured by recording a motor evoked potential (MEP) at the muscle level represented at the stimulated region level. Any increase or decrease in AMP amplitude, which persists after the end of TMS repetitive stimulation, indicates that there have been changes in the cortical, LTP or depression (LTD).
locomotion and posture | up to 3 years
  Stabilometric Platform
locomotion and posture | up to 3 years
  Gait Analysis
deglutition | up to 3 years
  Ectrophysiological and the Fibroendoscopic Deglutition Study
Cognition | up to 3 years
  ad-hoc tasks

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker R, McGinley JL, Schwartz MH, Beynon S, Rozumalski A, Graham HK, Tirosh O. The gait profile score and movement analysis profile. Gait Posture. 2009 Oct;30(3):265-9. doi: 10.1016/j.gaitpost.2009.05.020. Epub 2009 Jul 24. PMID 19632117
- [Background] Barkhof F. The clinico-radiological paradox in multiple sclerosis revisited. Curr Opin Neurol. 2002 Jun;15(3):239-45. doi: 10.1097/00019052-200206000-00003. PMID 12045719
- [Background] Bartlett TE, Wang YT. The intersections of NMDAR-dependent synaptic plasticity and cell survival. Neuropharmacology. 2013 Nov;74:59-68. doi: 10.1016/j.neuropharm.2013.01.012. Epub 2013 Jan 25. PMID 23357336
- [Background] Bliss TV, Lomo T. Long-lasting potentiation of synaptic transmission in the dentate area of the anaesthetized rabbit following stimulation of the perforant path. J Physiol. 1973 Jul;232(2):331-56. doi: 10.1113/jphysiol.1973.sp010273. PMID 4727084
- [Background] Nogueira LA, Teixeira L, Sabino P, Filho HA, Alvarenga RM, Thuler LC. Gait characteristics of multiple sclerosis patients in the absence of clinical disability. Disabil Rehabil. 2013 Aug;35(17):1472-8. doi: 10.3109/09638288.2012.738760. PMID 23869824
- [Background] Centonze D, Koch G, Versace V, Mori F, Rossi S, Brusa L, Grossi K, Torelli F, Prosperetti C, Cervellino A, Marfia GA, Stanzione P, Marciani MG, Boffa L, Bernardi G. Repetitive transcranial magnetic stimulation of the motor cortex ameliorates spasticity in multiple sclerosis. Neurology. 2007 Mar 27;68(13):1045-50. doi: 10.1212/01.wnl.0000257818.16952.62. PMID 17389310
- [Background] Centonze D, Rossi S, Tortiglione A, Picconi B, Prosperetti C, De Chiara V, Bernardi G, Calabresi P. Synaptic plasticity during recovery from permanent occlusion of the middle cerebral artery. Neurobiol Dis. 2007 Jul;27(1):44-53. doi: 10.1016/j.nbd.2007.03.012. Epub 2007 Apr 5. PMID 17490888
- [Background] Mori F, Rossi S, Piccinin S, Motta C, Mango D, Kusayanagi H, Bergami A, Studer V, Nicoletti CG, Buttari F, Barbieri F, Mercuri NB, Martino G, Furlan R, Nistico R, Centonze D. Synaptic plasticity and PDGF signaling defects underlie clinical progression in multiple sclerosis. J Neurosci. 2013 Dec 4;33(49):19112-9. doi: 10.1523/JNEUROSCI.2536-13.2013. PMID 24305808
- [Background] Chang PL, Isaacs KR, Greenough WT. Synapse formation occurs in association with the induction of long-term potentiation in two-year-old rat hippocampus in vitro. Neurobiol Aging. 1991 Sep-Oct;12(5):517-22. doi: 10.1016/0197-4580(91)90082-u. PMID 1770987
- [Background] Chumney D, Nollinger K, Shesko K, Skop K, Spencer M, Newton RA. Ability of Functional Independence Measure to accurately predict functional outcome of stroke-specific population: systematic review. J Rehabil Res Dev. 2010;47(1):17-29. doi: 10.1682/jrrd.2009.08.0140. PMID 20437324
- [Background] Ramaker C, Marinus J, Stiggelbout AM, Van Hilten BJ. Systematic evaluation of rating scales for impairment and disability in Parkinson's disease. Mov Disord. 2002 Sep;17(5):867-76. doi: 10.1002/mds.10248. PMID 12360535
- [Background] Comber L, Galvin R, Coote S. Gait deficits in people with multiple sclerosis: A systematic review and meta-analysis. Gait Posture. 2017 Jan;51:25-35. doi: 10.1016/j.gaitpost.2016.09.026. Epub 2016 Sep 26. PMID 27693958
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2002 Apr 6;359(9313):1221-31. doi: 10.1016/S0140-6736(02)08220-X. PMID 11955556
- [Background] D'Aniello A, Di Fiore MM, Fisher GH, Milone A, Seleni A, D'Aniello S, Perna AF, Ingrosso D. Occurrence of D-aspartic acid and N-methyl-D-aspartic acid in rat neuroendocrine tissues and their role in the modulation of luteinizing hormone and growth hormone release. FASEB J. 2000 Apr;14(5):699-714. doi: 10.1096/fasebj.14.5.699. PMID 10744627
- [Background] Di Lazzaro V, Profice P, Pilato F, Capone F, Ranieri F, Pasqualetti P, Colosimo C, Pravata E, Cianfoni A, Dileone M. Motor cortex plasticity predicts recovery in acute stroke. Cereb Cortex. 2010 Jul;20(7):1523-8. doi: 10.1093/cercor/bhp216. Epub 2009 Oct 5. PMID 19805417
- [Background] Duncan ID, Brower A, Kondo Y, Curlee JF Jr, Schultz RD. Extensive remyelination of the CNS leads to functional recovery. Proc Natl Acad Sci U S A. 2009 Apr 21;106(16):6832-6. doi: 10.1073/pnas.0812500106. Epub 2009 Apr 2. PMID 19342494
- [Background] Errico F, Nistico R, Napolitano F, Mazzola C, Astone D, Pisapia T, Giustizieri M, D'Aniello A, Mercuri NB, Usiello A. Increased D-aspartate brain content rescues hippocampal age-related synaptic plasticity deterioration of mice. Neurobiol Aging. 2011 Dec;32(12):2229-43. doi: 10.1016/j.neurobiolaging.2010.01.002. Epub 2010 Jan 25. PMID 20097447
- [Background] Errico F, Nistico R, Palma G, Federici M, Affuso A, Brilli E, Topo E, Centonze D, Bernardi G, Bozzi Y, D'Aniello A, Di Lauro R, Mercuri NB, Usiello A. Increased levels of d-aspartate in the hippocampus enhance LTP but do not facilitate cognitive flexibility. Mol Cell Neurosci. 2008 Feb;37(2):236-46. doi: 10.1016/j.mcn.2007.09.012. Epub 2007 Oct 5. PMID 17981050
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522
- [Background] Irvine KA, Blakemore WF. Remyelination protects axons from demyelination-associated axon degeneration. Brain. 2008 Jun;131(Pt 6):1464-77. doi: 10.1093/brain/awn080. Epub 2008 May 18. PMID 18490361
- [Background] Kalron A, Nitzani D, Magalashvili D, Dolev M, Menascu S, Stern Y, Rosenblum U, Pasitselsky D, Frid L, Zeilig G, Barmatz C, Givon U, Achiron A. A personalized, intense physical rehabilitation program improves walking in people with multiple sclerosis presenting with different levels of disability: a retrospective cohort. BMC Neurol. 2015 Mar 4;15:21. doi: 10.1186/s12883-015-0281-9. PMID 25884887
- [Background] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Background] Lamprecht R, LeDoux J. Structural plasticity and memory. Nat Rev Neurosci. 2004 Jan;5(1):45-54. doi: 10.1038/nrn1301. No abstract available. PMID 14708003
- [Background] Li R, Huang FS, Abbas AK, Wigstrom H. Role of NMDA receptor subtypes in different forms of NMDA-dependent synaptic plasticity. BMC Neurosci. 2007 Jul 26;8:55. doi: 10.1186/1471-2202-8-55. PMID 17655746
- [Background] Malenka RC, Nicoll RA. NMDA-receptor-dependent synaptic plasticity: multiple forms and mechanisms. Trends Neurosci. 1993 Dec;16(12):521-7. doi: 10.1016/0166-2236(93)90197-t. PMID 7509523
- [Background] Maletic-Savatic M, Malinow R, Svoboda K. Rapid dendritic morphogenesis in CA1 hippocampal dendrites induced by synaptic activity. Science. 1999 Mar 19;283(5409):1923-7. doi: 10.1126/science.283.5409.1923. PMID 10082466
- [Background] Mattson MP. Neurotransmitters in the regulation of neuronal cytoarchitecture. Brain Res. 1988 Apr-Jun;472(2):179-212. doi: 10.1016/0165-0173(88)90020-3. PMID 2898278
- [Background] Molina-Luna K, Pekanovic A, Rohrich S, Hertler B, Schubring-Giese M, Rioult-Pedotti MS, Luft AR. Dopamine in motor cortex is necessary for skill learning and synaptic plasticity. PLoS One. 2009 Sep 17;4(9):e7082. doi: 10.1371/journal.pone.0007082. PMID 19759902
- [Background] Mori F, Codeca C, Kusayanagi H, Monteleone F, Boffa L, Rimano A, Bernardi G, Koch G, Centonze D. Effects of intermittent theta burst stimulation on spasticity in patients with multiple sclerosis. Eur J Neurol. 2010 Feb;17(2):295-300. doi: 10.1111/j.1468-1331.2009.02806.x. Epub 2009 Oct 23. PMID 19863647
- [Background] Mori F, Kusayanagi H, Nicoletti CG, Weiss S, Marciani MG, Centonze D. Cortical plasticity predicts recovery from relapse in multiple sclerosis. Mult Scler. 2014 Apr;20(4):451-7. doi: 10.1177/1352458513512541. Epub 2013 Nov 21. PMID 24263385
- [Background] Mostert S, Kesselring J. Effects of a short-term exercise training program on aerobic fitness, fatigue, health perception and activity level of subjects with multiple sclerosis. Mult Scler. 2002 Apr;8(2):161-8. doi: 10.1191/1352458502ms779oa. PMID 11990874
- [Background] Motl RW, McAuley E. Longitudinal analysis of physical activity and symptoms as predictors of change in functional limitations and disability in multiple sclerosis. Rehabil Psychol. 2009 May;54(2):204-10. doi: 10.1037/a0015770. PMID 19469611
- [Background] Ota N, Shi T, Sweedler JV. D-Aspartate acts as a signaling molecule in nervous and neuroendocrine systems. Amino Acids. 2012 Nov;43(5):1873-86. doi: 10.1007/s00726-012-1364-1. Epub 2012 Aug 8. PMID 22872108
- [Background] Patrikios P, Stadelmann C, Kutzelnigg A, Rauschka H, Schmidbauer M, Laursen H, Sorensen PS, Bruck W, Lucchinetti C, Lassmann H. Remyelination is extensive in a subset of multiple sclerosis patients. Brain. 2006 Dec;129(Pt 12):3165-72. doi: 10.1093/brain/awl217. Epub 2006 Aug 18. PMID 16921173
- [Background] Pau M, Coghe G, Corona F, Marrosu MG, Cocco E. Effect of spasticity on kinematics of gait and muscular activation in people with Multiple Sclerosis. J Neurol Sci. 2015 Nov 15;358(1-2):339-44. doi: 10.1016/j.jns.2015.09.352. Epub 2015 Sep 18. PMID 26409825
- [Background] Pau M, Coghe G, Atzeni C, Corona F, Pilloni G, Marrosu MG, Cocco E, Galli M. Novel characterization of gait impairments in people with multiple sclerosis by means of the gait profile score. J Neurol Sci. 2014 Oct 15;345(1-2):159-63. doi: 10.1016/j.jns.2014.07.032. Epub 2014 Jul 19. PMID 25073571
- [Background] Richards DA, Mateos JM, Hugel S, de Paola V, Caroni P, Gahwiler BH, McKinney RA. Glutamate induces the rapid formation of spine head protrusions in hippocampal slice cultures. Proc Natl Acad Sci U S A. 2005 Apr 26;102(17):6166-71. doi: 10.1073/pnas.0501881102. Epub 2005 Apr 14. PMID 15831587
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Schirmer L, Merkler D, Konig FB, Bruck W, Stadelmann C. Neuroaxonal regeneration is more pronounced in early multiple sclerosis than in traumatic brain injury lesions. Brain Pathol. 2013 Jan;23(1):2-12. doi: 10.1111/j.1750-3639.2012.00608.x. Epub 2012 Jun 25. PMID 22612622
- [Background] Shi SH, Hayashi Y, Petralia RS, Zaman SH, Wenthold RJ, Svoboda K, Malinow R. Rapid spine delivery and redistribution of AMPA receptors after synaptic NMDA receptor activation. Science. 1999 Jun 11;284(5421):1811-6. doi: 10.1126/science.284.5421.1811. PMID 10364548
- [Background] Singer BH, Gamelli AE, Fuller CL, Temme SJ, Parent JM, Murphy GG. Compensatory network changes in the dentate gyrus restore long-term potentiation following ablation of neurogenesis in young-adult mice. Proc Natl Acad Sci U S A. 2011 Mar 29;108(13):5437-42. doi: 10.1073/pnas.1015425108. Epub 2011 Mar 14. PMID 21402918
- [Background] Solari A, Filippini G, Mendozzi L, Ghezzi A, Cifani S, Barbieri E, Baldini S, Salmaggi A, Mantia LL, Farinotti M, Caputo D, Mosconi P. Validation of Italian multiple sclerosis quality of life 54 questionnaire. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):158-62. doi: 10.1136/jnnp.67.2.158. PMID 10406981
- [Background] Stuifbergen AK, Blozis SA, Harrison TC, Becker HA. Exercise, functional limitations, and quality of life: A longitudinal study of persons with multiple sclerosis. Arch Phys Med Rehabil. 2006 Jul;87(7):935-43. doi: 10.1016/j.apmr.2006.04.003. PMID 16813781
- [Background] Trapp BD, Ransohoff R, Rudick R. Axonal pathology in multiple sclerosis: relationship to neurologic disability. Curr Opin Neurol. 1999 Jun;12(3):295-302. doi: 10.1097/00019052-199906000-00008. PMID 10499174
- [Background] Tyc F, Boyadjian A. Plasticity of motor cortex induced by coordination and training. Clin Neurophysiol. 2011 Jan;122(1):153-62. doi: 10.1016/j.clinph.2010.05.022. Epub 2010 Jun 17. PMID 21168091
- [Background] Wolff JR, Joo F, Dames W. Plasticity in dendrites shown by continuous GABA administration in superior cervical ganglion of adult rat. Nature. 1978 Jul 6;274(5666):72-4. doi: 10.1038/274072a0. No abstract available. PMID 661998
- [Background] Wolff JR, Missler M. Synaptic remodelling and elimination as integral processes of synaptogenesis. APMIS Suppl. 1993;40:9-23. PMID 8311996
- [Background] Yaka R, Biegon A, Grigoriadis N, Simeonidou C, Grigoriadis S, Alexandrovich AG, Matzner H, Schumann J, Trembovler V, Tsenter J, Shohami E. D-cycloserine improves functional recovery and reinstates long-term potentiation (LTP) in a mouse model of closed head injury. FASEB J. 2007 Jul;21(9):2033-41. doi: 10.1096/fj.06-7856com. Epub 2007 Mar 9. PMID 17351125
- [Background] Zepeda A, Aguilar-Arredondo A, Michel G, Ramos-Languren LE, Escobar ML, Arias C. Functional recovery of the dentate gyrus after a focal lesion is accompanied by structural reorganization in the adult rat. Brain Struct Funct. 2013 Mar;218(2):437-53. doi: 10.1007/s00429-012-0407-4. Epub 2012 Apr 6. PMID 22481229
- [Background] Ziemann U, Ilic TV, Pauli C, Meintzschel F, Ruge D. Learning modifies subsequent induction of long-term potentiation-like and long-term depression-like plasticity in human motor cortex. J Neurosci. 2004 Feb 18;24(7):1666-72. doi: 10.1523/JNEUROSCI.5016-03.2004. PMID 14973238